CLINICAL TRIAL: NCT06164561
Title: 18F-FAPI PET/MRI Imaging in the Diagnosis and Monitoring of Therapeutic Effect of Myelofibrosis: a Prospective Observational Study.
Brief Title: 18F-FAPI PET/MRI Imaging in Myelofibrosis: a Prospective Observational Study.
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Zhejiang Provincial Tongde Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Zhejiang Cancer Hospital (Other); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); First People's Hospital of Hangzhou (Other); Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IIT20230329B-R3
Record Dates: First submitted 2023-11-23; First posted 2023-12-11 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-02

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study intends to use a prospective, observational, self-controlled, multi-center study design to evaluate the feasibility and diagnostic efficacy of 18F-FDG PET/CT and 18F-FAPI PET/MRI imaging for the evaluation of systemic fibrosis in MF patients based on the results of bone marrow pathological biopsy, and to analyze the relationship between imaging results and clinical prognosis.

DETAILED DESCRIPTION:
Myelofibrosis (MF) is a pathological process characterized by dysplasia of bone marrow fibrous tissue, clonal proliferation of potential stem cells, inflammatory changes in the bone marrow microenvironment, and extramedullary hematopoiesis. Bone marrow histopathology is the gold standard for diagnosis, but because of the invasive nature of the puncture, repeated examination is not possible to dynamically monitor the disease process. In addition, due to the focal nature of puncture biopsy, it can not accurately reflect the systemic disease. 18F-FDG PET/CT provides visual assessment of MF, but its diagnostic effectiveness decreases as MF progresses. 18F-FAPI PET/MRI characterizes fiber activation processes in a variety of diseases. This study intends to use a prospective, observational, self-controlled, multi-center study design to evaluate the feasibility and diagnostic efficacy of 18F-FDG PET/CT and 18F-FAPI PET/MRI imaging for the evaluation of systemic fibrosis in MF patients based on the results of bone marrow pathological biopsy, and to analyze the relationship between imaging results and clinical prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary myelofibrosis or myelofibrosis secondary to myeloid tumors were diagnosed according to the diagnostic criteria of who 2022.
* Stable vital signs, ECOG score ≥ 2 points, tolerate and cooperate to complete 18F-FDG PET/CT and 18F-FAPI PET/MRI examination.
* The interval between imaging ,hematologic, cytogenetic and pathology was < 2 weeks.
* Willing to accept 18F-FDG PET/CT and 18F-FAPI PET/MRI , sign the informed consent.

Exclusion Criteria:

* Inability or unwillingness to provide informed consent.
* Other malignancies, autoimmune diseases, or chronic active infections were diagnosed within 1 year before the diagnosis of myelofibrosis.
* Current infection was present within 1 week before PET examination.
* Pregnant or lactation.
* Unable to follow protocol to complete follow-up.
* Have received glucocorticoid therapy within 2 weeks before PET imaging examination.
* Using granulocyte colony-stimulating factor (G-CSF) within 4 weeks prior to PET imaging.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: myelofibrosis
Sampling Method: Non-Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic efficiency of 18F-FAPI PET/MRI imaging in myelofibrosis | through study completion, an average of 2 years
  The diagnostic efficacy of 18F-FAPI PET/MRI in myelofibrosis was evaluated by visual scoring. The pattern of 18F-FAPI accumulation was analyzed on maximum-intensity projection images for each patient, and the extent of 18F-FAPI accumulation was graded on a 5-point scale（0-4） to assess changes in the extent of bone marrow involvement .The higher of the score, maybe the more severe in the myelofibrosis.The changes in diagnostic efficacy of 18F-FAPI PET/MRI imaging in myelofibrosis were compared with the gold standard of bone marrow biopsy by Kappa analysis.

SECONDARY OUTCOMES:
Comparison of clinical prognosis between pathological and 18F-FAPI PET/MRI imaging diagnosis by Kappa analysis. | through study completion, an average of 2 years
  To compare the clinical prognosis between pathological diagnosis and 18F-FAPI PET/MRI diagnosis by Kappa analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Sun, MD，Ph.D, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided